CLINICAL TRIAL: NCT03635099
Title: Phase II Evaluation of Safety, Tolerability, and Efficacy of BI 730357 in Patients With Moderate-to-severe Plaque Psoriasis
Brief Title: This Study is Done in Patients With Plaque Psoriasis and Tests How Well They Tolerate BI 730357 and How Effective it is
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1407-0030; 2017-004659-21 (EudraCT Number)
Record Dates: First submitted 2018-08-15; First posted 2018-08-17 (Actual); Results first posted 2022-06-02 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-07

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Part I - Placebo (fasted) (Placebo Comparator): Part I - Placebo matching BI 730357 taken orally once daily as a film-coated tablet in the morning while fasted for 12 weeks in period 1 followed by the same treatment for 12 weeks in period 2 (total treatment period of 24 weeks). Participants who failed to achieve a Psoriasis Area Severity Index score (PASI) 75 response at Week 12 were switched to a 200 mg dose, participants switching dose were imputed as failure for records after week 12, under original randomized treatment arm.
  Interventions: Drug: Placebo (fasted)
- Part I - BI 25 mg (fasted) (Experimental): Part I - 25 milligram (mg) BI 730357 taken orally once daily as a film-coated tablet in the morning while fasted for 12 weeks in period 1 followed by the same treatment for 12 weeks in period 2 (total treatment period of 24 weeks). Participants who failed to achieve a Psoriasis Area Severity Index score (PASI) 50 response at Week 12 were switched to a 50 mg dose, participants switching dose were imputed as failure for records after week 12, under original randomized treatment arm.
  Interventions: Drug: BI 25 mg (fasted)
- Part I - BI 50 mg (fasted) (Experimental): Part I - 50 milligram (mg) BI 730357 taken orally once daily as a film-coated tablet in the morning while fasted for 12 weeks in period 1 followed by the same treatment for 12 weeks in period 2 (total treatment period of 24 weeks). Participants who failed to achieve a Psoriasis Area Severity Index score (PASI) 50 response at Week 12 were switched to a 100 mg dose, participants switching dose were imputed as failure for records after week 12, under original randomized treatment arm.
  Interventions: Drug: BI 50 mg (fasted)
- Part I - BI 100 mg (fasted) (Experimental): Part I - 100 milligram (mg) BI 730357 taken orally once daily as a film-coated tablet in the morning while fasted for 12 weeks in period 1 followed by the same treatment for 12 weeks in period 2 (total treatment period of 24 weeks). Participants who failed to achieve a Psoriasis Area Severity Index score (PASI) 50 response at Week 12 were switched to a 200 mg dose, participants switching dose were imputed as failure for records after week 12, under original randomized treatment arm.
  Interventions: Drug: BI 100 mg (fasted)
- Part I - BI 200 mg (fasted) (Experimental): Part I - 200 milligram (mg) BI 730357 taken orally once daily as a film-coated tablet in the morning while fasted for 12 weeks in period 1 followed by the same treatment for 12 weeks in period 2 (total treatment period of 24 weeks).
  Interventions: Drug: BI 200 mg (fasted)
- Part II - Placebo (fed) (Placebo Comparator): Part II - 4 film-coated tablets of matching Placebo were taken orally in the morning with a meal and 2 film-coated tablets of matching Placebo were taken orally in the evening with a meal for 12 weeks.
  Interventions: Drug: Placebo (fed)
- Part II - BI 400 mg once daily (fed) (Experimental): Part II - 4 film-coated tablets of 100 milligram (mg) BI 730357 (400 mg in total) were taken orally in the morning with a meal and 2 film-coated tablets of matching Placebo were taken orally in the evening with a meal for 12 weeks.
  Interventions: Drug: BI 400 mg once daily (fed)
- Part II - BI 200 mg twice daily, 400 mg total (fed) (Experimental): Part II - 2 film-coated tablets of 100 milligram (mg) BI 730357 were taken orally with a meal in the morning and evening (twice daily; total daily dosage: 400 mg) for 12 weeks.
  Interventions: Drug: BI 200 mg twice daily, 400 mg total (fed)

INTERVENTIONS:
Drug: Placebo (fasted) — Placebo matching BI 730357 taken orally once daily as a film-coated tablet in the morning while fasted for 12 weeks in period 1 followed by the same treatment for 12 weeks in period 2 (total treatment period of 24 weeks).
  Arms: Part I - Placebo (fasted)
Drug: BI 25 mg (fasted) — 25 milligram (mg) BI 730357 taken orally once daily as a film-coated tablet in the morning while fasted for 12 weeks in period 1 followed by the same treatment for 12 weeks in period 2 (total treatment period of 24 weeks).
  Arms: Part I - BI 25 mg (fasted)
Drug: BI 50 mg (fasted) — 50 milligram (mg) BI 730357 taken orally once daily as a film-coated tablet in the morning while fasted for 12 weeks in period 1 followed by the same treatment for 12 weeks in period 2 (total treatment period of 24 weeks).
  Arms: Part I - BI 50 mg (fasted)
Drug: BI 100 mg (fasted) — 100 milligram (mg) BI 730357 taken orally once daily as a film-coated tablet in the morning while fasted for 12 weeks in period 1 followed by the same treatment for 12 weeks in period 2 (total treatment period of 24 weeks).
  Arms: Part I - BI 100 mg (fasted)
Drug: BI 200 mg (fasted) — 200 milligram (mg) BI 730357 taken orally once daily as a film-coated tablet in the morning while fasted for 12 weeks in period 1 followed by the same treatment for 12 weeks in period 2 (total treatment period of 24 weeks).
  Arms: Part I - BI 200 mg (fasted)
Drug: Placebo (fed) — 4 film-coated tablets of matching Placebo were taken orally in the morning with a meal and 2 film-coated tablets of matching Placebo were taken orally in the evening with a meal for 12 weeks.
  Arms: Part II - Placebo (fed)
Drug: BI 400 mg once daily (fed) — 4 film-coated tablets of 100 milligram (mg) BI 730357 (400 mg in total) were taken orally in the morning with a meal and 2 film-coated tablets of matching Placebo were taken orally in the evening with a meal for 12 weeks.
  Arms: Part II - BI 400 mg once daily (fed)
Drug: BI 200 mg twice daily, 400 mg total (fed) — 2 film-coated tablets of 100 milligram (mg) BI 730357 were taken orally with a meal in the morning and evening (twice daily; total daily dosage: 400 mg) for 12 weeks.
  Arms: Part II - BI 200 mg twice daily, 400 mg total (fed)

SUMMARY:
The primary objective is based on Week 12 co-primary endpoints of PASI (Psoriasis Area and Severity Index) 75 and sPGA (Static Physician's Global Assessment) 0/1, and overall safety Secondary objectives of Part 1 are to evaluate the efficacy and safety of BI 730357 through 24 weeks of treatment

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients. Woman Of Childbearing Potential (WoCBP) must be ready and able to use highly effective methods of birth control per International Conference on Harmonisation (ICH) M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly from date of screening until 4 weeks after last treatment in this trial. A list of contraception methods meeting these criteria is provided in the patient information.
* Age 18 to 75 years (both inclusive) at screening
* BMI < 35 kg/m2 at screening
* Diagnosis of chronic plaque psoriasis (with or without psoriatic arthritis) for at least 6 months before the first administration of study drug. Duration of diagnosis may be reported by the patient
* Patients must be candidates for systemic PsO therapy.Moderate-to-severe plaque psoriasis:

  * BSA ≥10% and
  * PASI ≥12 and
  * sPGA moderate or severe
* Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial

Exclusion Criteria:

* Nonplaque forms of PsO (including guttate, erythrodermic, or pustular), current druginduced PsO (including a new onset or exacerbation of PsO from, e.g., beta blockers, calcium channel blockers, lithium), active ongoing inflammatory diseases (including but not limited to Inflammatory bowel disease (IBD)) other than PsO that might confound trial evaluations
* Previous enrolment in this trial or previous exposure to BI 730357.
* Current enrollment in another investigational device or drug trial, or is less than 30 days (from randomisation) since ending another investigational device or drug trial(s), or receipt of other investigational treatment(s).
* Use of

  * any biologic agent within 12 weeks, or
  * any anti IL-23 biologic agent within 24 weeks prior to randomisation, or
  * systemic anti-psoriatic medications or phototherapy within 4 weeks prior to randomisation, or
  * topical anti-psoriasis medications within 2 weeks prior to randomisation
* Receipt of a live vaccination within 12 weeks prior to randomisation (visit 2), or any plan to receive a live vaccination during the conduct of this trial
* Patients who must or wish to continue the intake of restricted medications or any drug considered likely to interfere with the safe conduct of the trial
* Patients not expected to comply with the protocol requirements or not expected to complete the trial as scheduled.
* Chronic alcohol or drug abuse or any condition that, in the investigator's opinion, makes the patient an unreliable trial participant or unlikely to complete the trial.
* Major surgery (major according to the investigator's assessment) performed within 12 weeks prior to randomisation or planned within 12 months after screening, e.g., hip replacement
* Women who are pregnant, nursing, or who plan to become pregnant while in the trial
* Any documented active or suspected malignancy or history of malignancy within 5 years prior to screening, except appropriately treated basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ carcinoma of uterine cervix
* Relevant chronic or acute infections including human immunodeficiency virus (HIV), viral hepatitis, candidiasis and tuberculosis. A patient can be re-screened if the patient was treated and is cured from the acute infection.
* Evidence of a current or previous disease (including known or suspected IBD, and cardiovascular disease), or medical finding that in the opinion of the investigator is clinically significant and would make the study participant unreliable to adhere to the protocol or to complete the trial, compromise the safety of the patient, or compromise the quality of the data.
* Any suicidal ideation, including grade 4 or 5 in the Columbia Suicide Severity Rating Scale (CSSRS) in the past 3 months (i.e., active suicidal thought with intent but without specific plan, or active suicidal thought with plan and intent).
* Unwillingness to adhere to the rules of UV-light protection
* Further exclusion criteria apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2021-05-06 (Actual); Study Completion 2021-05-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (34):
- United States (16):
  - Total Skin and Beauty Dermatology Center, PC, Birmingham, Alabama
  - Dermatology Research Associates, Los Angeles, California
  - Southern California Dermatology Inc., Santa Ana, California
  - Hamilton Research, Alpharetta, Georgia
  - Advanced Medical Research PC, Sandy Springs, Georgia
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - The Psoriasis Treatment Center of Central New Jersey, East Windsor, New Jersey
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Synexus, Cincinnati, Ohio
  - Clinical Partners, LLC, Johnston, Rhode Island
  - Clinical Research Center of the Carolinas, Charleston, South Carolina
  - Health Concepts, Rapid City, South Dakota
  - Menter Dermatology Research Institute, Dallas, Texas
  - Center for Clinical Studies, Houston, Texas
  - Center for Clinical Studies, Webster, Texas
  - Virginia Clinical Research, Inc., Norfolk, Virginia
- Canada (11):
  - Dr Chih-ho Hong Medical Inc, Surrey, British Columbia
  - Enverus Medical Research, Surrey, British Columbia
  - Dr. Irina Turchin PC Inc., Fredericton, New Brunswick
  - The Guenther Dermatology Research Centre, London, Ontario
  - DermEdge Research Inc., Mississauga, Ontario
  - North Bay Dermatology Centre, North Bay, Ontario
  - The Centre for Clinical Trials, Oakville, Ontario
  - SKiN Centre for Dermatology, Peterborough, Ontario
  - The Centre for Dermatology, Richmond Hill, Ontario
  - K. Papp Clinical Research Inc., Waterloo, Ontario
  - XLR8 Medical Research Inc., Windsor, Ontario
- Germany (7):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Studienzentrum im Jahrhunderthaus, Bochum
  - Universitätsklinikum Frankfurt, Frankfurt am Main
  - TFS Trial Form Support GmbH, Hamburg
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum Schleswig-Holstein, Campus Lübeck, Lübeck
  - Universitätsklinikum Münster, Münster

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed and the primary manuscript is accepted for publishing, researchers can use this following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Also, Researchers can use the following link https://www.mystudywindow.com/msw/datasharing to find information in order to request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
  The data shared are the raw clinical study data sets.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by both the independent review panel and the sponsor, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a 'Data Sharing Agreement'.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] Gooderham MJ, Mrowietz U, Kadus W, Drda K, Gu H, Vangerow H, Flack M, Korell J, Sofen H, Papp KA. Phase II Randomized Trial of BI 730357, an Oral RORgammat Inhibitor, for Moderate-to-Severe Plaque Psoriasis. J Invest Dermatol. 2025 Aug;145(8):1969-1978.e14. doi: 10.1016/j.jid.2024.12.025. Epub 2025 Jan 21. PMID 39848568
- [Derived] Ooi QX, Kristoffersson A, Korell J, Flack M, L Plan E, Weber B. Bounded integer model-based analysis of psoriasis area and severity index in patients with moderate-to-severe plaque psoriasis receiving BI 730357. CPT Pharmacometrics Syst Pharmacol. 2023 Jun;12(6):758-769. doi: 10.1002/psp4.12948. Epub 2023 May 1. PMID 36919398
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was a 2-part, randomised, placebo-controlled, double-blind, parallel-group, dose-ranging trial to investigate the efficacy, safety, and tolerability of different dose regimens of BI 730357 in patients with moderate-to-severe plaque psoriasis.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Period: Period 1
Arm/Group | Part I - Placebo (Fasted) | Part I - BI 25 mg (Fasted) | Part I - BI 50 mg (Fasted) | Part I - BI 100 mg (Fasted) | Part I - BI 200 mg (Fasted) | Part II - Placebo (Fed) | Part II - BI 400 mg Once Daily (Fed) | Part II - BI 200 mg Twice Daily, 400 mg Total (Fed)
Started | 20 | 40 | 39 | 39 | 40 | 10 | 44 | 42
Full Analysis Set (FAS) | 20 | 40 | 39 | 39 | 40 | 10 | 43 | 42
Completed (Completed period 1: completed 12 weeks of treatment.) | 16 | 37 | 31 | 34 | 37 | 9 | 40 | 40
Not Completed | 4 | 3 | 8 | 5 | 3 | 1 | 4 | 2
Not completed — Adverse Event | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 2 | 1 | 0 | 1 | 2
Not completed — Withdrawal by Subject | 3 | 3 | 5 | 2 | 2 | 0 | 3 | 0
Not completed — History of suicidal ideation | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — pursue other treatment options | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Period: Not Eligible for Period 2
Arm/Group | Part I - Placebo (Fasted) | Part I - BI 25 mg (Fasted) | Part I - BI 50 mg (Fasted) | Part I - BI 100 mg (Fasted) | Part I - BI 200 mg (Fasted) | Part II - Placebo (Fed) | Part II - BI 400 mg Once Daily (Fed) | Part II - BI 200 mg Twice Daily, 400 mg Total (Fed)
Started | 16 | 37 | 31 | 34 | 37 | 9 | 40 | 40
Completed (Completed subjects moved to period 2. Not completed did not move to period 2.) | 15 | 37 | 31 | 33 | 37 | 0 | 0 | 0
Not Completed | 1 | 0 | 0 | 1 | 0 | 9 | 40 | 40
Not completed — Pregnancy | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Part II subjects did not have a period 2. | 0 | 0 | 0 | 0 | 0 | 9 | 40 | 40
Period: Eligible for Period 2
Arm/Group | Part I - Placebo (Fasted) | Part I - BI 25 mg (Fasted) | Part I - BI 50 mg (Fasted) | Part I - BI 100 mg (Fasted) | Part I - BI 200 mg (Fasted) | Part II - Placebo (Fed) | Part II - BI 400 mg Once Daily (Fed) | Part II - BI 200 mg Twice Daily, 400 mg Total (Fed)
Started | 15 | 37 | 31 | 33 | 37 | 0 | 0 | 0
Switching Patients (Non-responding patients in dose groups were switched at the end of period 1 to a higher dose group.) | 15 (Switched to the 'BI 200 mg' dose group.) | 35 (Switched to the 'BI 50 mg' dose group.) | 21 (Switched to the 'BI 100 mg' dose group.) | 25 (Switched to the 'BI 200 mg' dose group.) | 0 | 0 | 0 | 0
Non Switching Patients (Patients stayed in initially randomized treatment group.) | 0 | 2 | 10 | 8 | 37 | 0 | 0 | 0
Completed | 0 | 2 | 10 | 8 | 37 | 0 | 0 | 0
Not Completed | 15 | 35 | 21 | 25 | 0 | 0 | 0 | 0
Not completed — Switch to higher dose at end of period 1 | 15 | 35 | 21 | 25 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Part I - Placebo (Fasted) | Part I - BI 25 mg (Fasted) | Part I - BI 50 mg (Fasted) | Part I - BI 100 mg (Fasted) | Part I - BI 200 mg (Fasted) | Part II - Placebo (Fed) | Part II - BI 400 mg Once Daily (Fed) | Part II - BI 200 mg Twice Daily, 400 mg Total (Fed)
Started | 0 | 2 | 45 (Combination of period 1 dose groups: "BI 50 mg" and switched patients from dose Group "BI 25 mg") | 29 (Combination of period 1 dose groups: "BI 100 mg" and switched patients from dose Group "BI 50 mg") | 77 (Combination of period 1: "BI 200mg", switched patients from dose Group "BI 100 mg" and "Placebo".) | 0 | 0 | 0
Completed | 0 | 2 | 36 | 25 | 65 | 0 | 0 | 0
Not Completed | 0 | 0 | 9 | 4 | 12 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 4 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 7 | 4 | 7 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): The FAS includes all patients who received at least 1 dose of trial medication and provided baseline and at least 1 post-randomisation measurement of Psoriasis Area Severity Index (PASI).
Groups:
- Total: Total of all reporting groups
Arm/Group | Part I - Placebo (Fasted) | Part I - BI 25 mg (Fasted) | Part I - BI 50 mg (Fasted) | Part I - BI 100 mg (Fasted) | Part I - BI 200 mg (Fasted) | Part II - Placebo (Fed) | Part II - BI 400 mg Once Daily (Fed) | Part II - BI 200 mg Twice Daily, 400 mg Total (Fed) | Total
Number analyzed (Participants) | 20 | 40 | 39 | 39 | 40 | 10 | 43 | 42 | 273
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.1 (14.7) | 47.2 (13.7) | 46.3 (15.1) | 47.6 (14.4) | 43.8 (13.1) | 51.6 (16.3) | 44.1 (14.7) | 43.7 (11.5) | 45.8 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 15 | 14 | 12 | 14 | 3 | 6 | 16 | 84
  Male | 16 | 25 | 25 | 27 | 26 | 7 | 37 | 26 | 189
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 9 | 8 | 10 | 7 | 2 | 11 | 11 | 62
  Not Hispanic or Latino | 16 | 31 | 31 | 29 | 33 | 8 | 32 | 31 | 211
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 1 | 2 | 3 | 1 | 1 | 5 | 4 | 20
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Black or African American | 1 | 2 | 3 | 2 | 2 | 1 | 5 | 4 | 20
  White | 16 | 37 | 33 | 34 | 37 | 7 | 33 | 33 | 230
  More than one race | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Psoriasis Area Severity Index score (PASI) [Mean (Standard Deviation); unit: Score on scale] — The PASI is a tool which provides a numeric scoring for patients overall psoriasis disease state, ranging from 0 to 72. It is a linear combination of percent of surface area of skin that is affected and the severity of erythema, infiltration, and desquamation over four body regions. Higher scores indicating higher severity, while a score of 0 indicates no disease.
  Score on scale | 17.1 (5.2) | 17.4 (6.2) | 18.3 (4.8) | 18.6 (6.0) | 16.8 (6.6) | 17.8 (5.4) | 18.8 (7.1) | 17.9 (7.4) | 17.9 (6.3)
Static Physician's Global Assessment score (sPGA) [Count of Participants; unit: Participants] — The sPGA is a 5 point score (0 to 4) based on the physician's assessment of the average thickness, erythema, and scaling of all psoriatic lesions. A lower score indicates less body coverage, with 0 being clear , 1 almost clear, 2 mild, 3 moderate and 5 severe. Reported are the number of subjects with a moderate (dull to bright red coloration, clearly distinguishable to moderate thickening, moderate scaling) and severe (bright to deep dark red coloration, severe thickening with hard edges, severe coarse scaling covering almost all or all lesions) score.
  Participants
    Moderate | 16 | 35 | 29 | 34 | 30 | 7 | 34 | 34 | 219
    Severe | 4 | 5 | 10 | 5 | 10 | 3 | 9 | 8 | 54

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Achieved Psoriasis Area Severity Index Score (PASI) 75 at Week 12
Description: Number of patients who achieved Psoriasis Area Severity Index score (PASI) 75 at week 12. The PASI is a tool which provides a numeric scoring for patients overall psoriasis disease state, ranging from 0 to 72. It is a linear combination of percent of surface area of skin that is affected and the severity of erythema, infiltration, and desquamation over four body regions. Higher scores indicating higher severity, while a score of 0 indicates no disease.
  PASI 75 is based on the percent reduction from baseline, generally summarized as a dichotomous outcome based on achieving over an 75% reduction.
  No statistical comparisons were planned or carried out for Part 2 of the trial.
Time Frame: Assesment at week 12 of treatment
Population: Full Analysis Set (FAS): The FAS includes all patients who received at least 1 dose of trial medication and provided baseline and at least 1 post-randomisation measurement of Psoriasis Area Severity Index (PASI). Subjects with missing data for subsequent visits were included but those entries were imputed as failures.
Measure: Count of Participants; unit: Participants
Arm/Group | Part I - Placebo (Fasted) | Part I - BI 25 mg (Fasted) | Part I - BI 50 mg (Fasted) | Part I - BI 100 mg (Fasted) | Part I - BI 200 mg (Fasted) | Part II - Placebo (Fed) | Part II - BI 400 mg Once Daily (Fed) | Part II - BI 200 mg Twice Daily, 400 mg Total (Fed)
Number analyzed (Participants) | 20 | 40 | 39 | 39 | 40 | 10 | 43 | 42
Participants | 0 | 2 | 3 | 4 | 12 | 0 | 11 | 10
Statistical Analysis 1: Comparison: Part I - Placebo (Fasted) vs Part I - BI 25 mg (Fasted); Test type: Other; p = 0.3091, Chi-squared; Risk Difference (RD) = 5.0, 95% CI 2-sided [-1.8 to 11.8] — Statistics for the difference were calculated using unadjusted risk differences (BI dose group - Placebo)
Statistical Analysis 2: Comparison: Part I - Placebo (Fasted) vs Part I - BI 50 mg (Fasted); Test type: Other; p = 0.2030, Chi-squared; Risk Difference (RD) = 7.7, 95% CI 2-sided [-0.7 to 16.1] — Statistics for the difference were calculated using unadjusted risk differences (BI dose group - Placebo)
Statistical Analysis 3: Comparison: Part I - Placebo (Fasted) vs Part I - BI 100 mg (Fasted); Test type: Other; p = 0.1380, Chi-squared; Risk Difference (RD) = 10.3, 95% CI 2-sided [0.7 to 19.8] — Statistics for the difference were calculated using unadjusted risk differences (BI dose group - Placebo)
Statistical Analysis 4: Comparison: Part I - Placebo (Fasted) vs Part I - BI 200 mg (Fasted); Test type: Other; p = 0.0062, Chi-squared; Risk Difference (RD) = 30.0, 95% CI 2-sided [15.8 to 44.2] — Statistics for the difference were calculated using unadjusted risk differences (BI dose group - Placebo)
Statistical Analysis 5: Comparison: Part II - Placebo (Fed) vs Part II - BI 400 mg Once Daily (Fed); The 95% confidence interval for the unadjusted absolute difference in proportion (%) between active group and placebo group was estimated by Chi-square method. As pre-specified, no hypothesis testing was carried out for Part 2 of this trial and no p-values were provided; Test type: Other; Risk Difference (RD) = 25.6, 95% CI 2-sided [12.5 to 38.6] — Statistics for the difference were calculated using unadjusted risk differences (BI dose group - Placebo)
Statistical Analysis 6: Comparison: Part II - Placebo (Fed) vs Part II - BI 200 mg Twice Daily, 400 mg Total (Fed); [analysis description as in outcome 1, analysis 5]; Test type: Other; Risk Difference (RD) = 23.8, 95% CI 2-sided [10.9 to 36.7] — Statistics for the difference were calculated using unadjusted risk differences (BI dose group - Placebo)
Statistical Analysis 7: Comparison: Part I - Placebo (Fasted) vs Part I - BI 25 mg (Fasted) vs Part I - BI 50 mg (Fasted) vs Part I - BI 100 mg (Fasted) vs Part I - BI 200 mg (Fasted); Test type: Other — First the response rate of PASI 75 at week 12 for each dosage group was estimated by a logistic regression model including the fixed effect of treatment (categorical dose) and baseline PASI score as covariate was performed. The dose-response relationships were then tested using the Multiple Comparison Procedures and Modelling (MCP-Mod) approach based on the estimates from logistic regression; p = 0.0004, MCPMod Linear model fit. — The multiple comparison procedure was implemented using optimal contrast tests which control the family-wise type I error rate at one-sided α = 0.05
Statistical Analysis 8: Comparison: Part I - Placebo (Fasted) vs Part I - BI 25 mg (Fasted) vs Part I - BI 50 mg (Fasted) vs Part I - BI 100 mg (Fasted) vs Part I - BI 200 mg (Fasted); Test type: Other — [test comment as in outcome 1, analysis 7]; p = 0.0012, MCPMod Logistic model fit. — [p-value comment as in outcome 1, analysis 7]; Model assumption: 10% of the maximum effect is achieved at 25 mg and 80% of the maximum effect is achieved at 100 mg
Statistical Analysis 9: Comparison: Part I - Placebo (Fasted) vs Part I - BI 25 mg (Fasted) vs Part I - BI 50 mg (Fasted) vs Part I - BI 100 mg (Fasted) vs Part I - BI 200 mg (Fasted); Test type: Other — [test comment as in outcome 1, analysis 7]; p = 0.0008, MCPMod Emax1 model fit. — [p-value comment as in outcome 1, analysis 7]; Model assumption: 30% of the maximum effect is achieved at 50 mg
Statistical Analysis 10: Comparison: Part I - Placebo (Fasted) vs Part I - BI 25 mg (Fasted) vs Part I - BI 50 mg (Fasted) vs Part I - BI 100 mg (Fasted) vs Part I - BI 200 mg (Fasted); Test type: Other — [test comment as in outcome 1, analysis 7]; p = 0.0217, MCPMod Emax2 model fit. — [p-value comment as in outcome 1, analysis 7]; Model assumption: 80% of the maximum effect is achieved at 50 mg
Statistical Analysis 11: Comparison: Part I - Placebo (Fasted) vs Part I - BI 25 mg (Fasted) vs Part I - BI 50 mg (Fasted) vs Part I - BI 100 mg (Fasted) vs Part I - BI 200 mg (Fasted); Test type: Other — [test comment as in outcome 1, analysis 7]; p = 0.0004, MCPMod Exponential model fit. — [p-value comment as in outcome 1, analysis 7]; Model assumption: 5% of the maximum effect is achieved at 25 mg

2. Primary Outcome: Number of Patients Who Achieved a Static Physician's Global Assessment Score of 'Clear' or 'Almost Clear' (sPGA 0/1) at Week 12.
Description: Number of patients who achieved a static Physician's Global Assessment score of 'clear' or 'almost clear' (sPGA 0/1) at Week 12. The sPGA used in this trial is a 5 point score ranging from 0 to 4, based on the physician's assessment of the average thickness, erythema, and scaling of all psoriatic lesions. The assessment is considered "static" which refers to the patients disease state at the time of the assessments, without comparison to any of the subject's previous disease states, whether at Baseline or at a previous visit. A lower score indicates less body coverage, with 0 being clear and 1 being almost clear.
  No statistical comparisons were planned or carried out for Part 2 of the trial.
Time Frame: Assesment at week 12 of treatment
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part I - Placebo (Fasted) | Part I - BI 25 mg (Fasted) | Part I - BI 50 mg (Fasted) | Part I - BI 100 mg (Fasted) | Part I - BI 200 mg (Fasted) | Part II - Placebo (Fed) | Part II - BI 400 mg Once Daily (Fed) | Part II - BI 200 mg Twice Daily, 400 mg Total (Fed)
Number analyzed (Participants) | 20 | 40 | 39 | 39 | 40 | 10 | 43 | 42
Participants | 0 | 1 | 3 | 2 | 11 | 0 | 11 | 10
Statistical Analysis 1: Comparison: Part I - Placebo (Fasted) vs Part I - BI 25 mg (Fasted); Test type: Other; p = 0.4758, Chi-squared; Risk Difference (RD) = 2.5, 95% CI 2-sided [-2.3 to 7.3] — Statistics for the difference were calculated using unadjusted risk differences (BI dose group - Placebo)
Statistical Analysis 2: Comparison: Part I - Placebo (Fasted) vs Part I - BI 50 mg (Fasted); Test type: Other; p = 0.2030, Chi-squared; Risk Difference (RD) = 7.7, 95% CI 2-sided [-0.7 to 16.1] — Statistics for the difference were calculated using unadjusted risk differences (BI dose group - Placebo)
Statistical Analysis 3: Comparison: Part I - Placebo (Fasted) vs Part I - BI 100 mg (Fasted); Test type: Other; p = 0.3028, Chi-squared; Risk Difference (RD) = 5.1, 95% CI 2-sided [-1.8 to 12.1] — Statistics for the difference were calculated using unadjusted risk differences (BI dose group - Placebo)
Statistical Analysis 4: Comparison: Part I - Placebo (Fasted) vs Part I - BI 200 mg (Fasted); Test type: Other; p = 0.0095, Chi-squared; Risk Difference (RD) = 27.5, 95% CI 2-sided [13.7 to 41.3] — Statistics for the difference were calculated using unadjusted risk differences (BI dose group - Placebo)
Statistical Analysis 5: Comparison: Part I - Placebo (Fasted) vs Part I - BI 25 mg (Fasted) vs Part I - BI 50 mg (Fasted) vs Part I - BI 100 mg (Fasted) vs Part I - BI 200 mg (Fasted); Test type: Other — First the response rate of sPGA 0/1 at week 12 for each dosage group was estimated by a logistic regression model including the fixed effect of treatment (categorical dose) and baseline sPGA score as covariate was performed. The dose-response relationships were then tested using the Multiple Comparison Procedures and Modelling (MCP-Mod) approach based on the estimates from logistic regression; p = 0.0007, MCPMod Linear model fit. — [p-value comment as in outcome 1, analysis 7]
Statistical Analysis 6: Comparison: Part I - Placebo (Fasted) vs Part I - BI 25 mg (Fasted) vs Part I - BI 50 mg (Fasted) vs Part I - BI 100 mg (Fasted) vs Part I - BI 200 mg (Fasted); Test type: Other — [test comment as in outcome 2, analysis 5]; p = 0.0023, MCPMod Logistic model fit. — [p-value comment as in outcome 1, analysis 7]; Model assumption: 10% of the maximum effect is achieved at 25 mg and 80% of the maximum effect is achieved at 100 mg
Statistical Analysis 7: Comparison: Part I - Placebo (Fasted) vs Part I - BI 25 mg (Fasted) vs Part I - BI 50 mg (Fasted) vs Part I - BI 100 mg (Fasted) vs Part I - BI 200 mg (Fasted); Test type: Other — [test comment as in outcome 2, analysis 5]; p = 0.0018, MCPMod Emax1 model fit. — [p-value comment as in outcome 1, analysis 7]; Model assumption: 30% of the maximum effect is achieved at 50 mg
Statistical Analysis 8: Comparison: Part I - Placebo (Fasted) vs Part I - BI 25 mg (Fasted) vs Part I - BI 50 mg (Fasted) vs Part I - BI 100 mg (Fasted) vs Part I - BI 200 mg (Fasted); Test type: Other — [test comment as in outcome 2, analysis 5]; p = 0.0386, MCPMod Emax2 model fit. — [p-value comment as in outcome 1, analysis 7]; Model assumption: 80% of the maximum effect is achieved at 50 mg
Statistical Analysis 9: Comparison: Part I - Placebo (Fasted) vs Part I - BI 25 mg (Fasted) vs Part I - BI 50 mg (Fasted) vs Part I - BI 100 mg (Fasted) vs Part I - BI 200 mg (Fasted); Test type: Other — [test comment as in outcome 2, analysis 5]; p = 0.0004, MCPMod Exponential model fit. — [p-value comment as in outcome 1, analysis 7]; Model assumption: 5% of the maximum effect is achieved at 25 mg

3. Secondary Outcome: Number of Patients Who Achieved Psoriasis Area Severity Index Score (PASI) 50 at Week 12
Description: Number of patients who achieved Psoriasis Area Severity Index score (PASI) 50 at week 12. The PASI is a tool which provides a numeric scoring for patients overall psoriasis disease state, ranging from 0 to 72. It is a linear combination of percent of surface area of skin that is affected and the severity of erythema, infiltration, and desquamation over four body regions. Higher scores indicating higher severity, while a score of 0 indicates no disease.
  PASI 50 is based on the percent reduction from baseline, generally summarized as a dichotomous outcome based on achieving over an 50% reduction.
  No hypothesis testing was planned or carried out for Part II.
Time Frame: Assesment at week 12 of treatment
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part I - Placebo (Fasted) | Part I - BI 25 mg (Fasted) | Part I - BI 50 mg (Fasted) | Part I - BI 100 mg (Fasted) | Part I - BI 200 mg (Fasted) | Part II - Placebo (Fed) | Part II - BI 400 mg Once Daily (Fed) | Part II - BI 200 mg Twice Daily, 400 mg Total (Fed)
Number analyzed (Participants) | 20 | 40 | 39 | 39 | 40 | 10 | 43 | 42
Participants | 1 | 2 | 10 | 8 | 20 | 1 | 24 | 19
Statistical Analysis 1: Comparison: Part I - Placebo (Fasted) vs Part I - BI 25 mg (Fasted); Test type: Other; p = 1.0000, Chi-squared; Risk Difference (RD) = 0.0, 95% CI 2-sided [-11.7 to 11.7] — Statistics for the difference were calculated using unadjusted risk differences (BI dose group - Placebo)
Statistical Analysis 2: Comparison: Part I - Placebo (Fasted) vs Part I - BI 50 mg (Fasted); Test type: Other; p = 0.0540, Chi-squared; Risk Difference (RD) = 20.6, 95% CI 2-sided [3.9 to 37.3] — Statistics for the difference were calculated using unadjusted risk differences (BI dose group - Placebo)
Statistical Analysis 3: Comparison: Part I - Placebo (Fasted) vs Part I - BI 100 mg (Fasted); Test type: Other; p = 0.1167, Chi-squared; Risk Difference (RD) = 15.5, 95% CI 2-sided [-0.4 to 31.4] — Statistics for the difference were calculated using unadjusted risk differences (BI dose group - Placebo)
Statistical Analysis 4: Comparison: Part I - Placebo (Fasted) vs Part I - BI 200 mg (Fasted); Test type: Other; p = 0.0006, Chi-squared; Risk Difference (RD) = 45.0, 95% CI 2-sided [26.8 to 63.2] — Statistics for the difference were calculated using unadjusted risk differences (BI dose group - Placebo)
Statistical Analysis 5: Comparison: Part II - Placebo (Fed) vs Part II - BI 400 mg Once Daily (Fed); [analysis description as in outcome 1, analysis 5]; Test type: Other; Risk Difference (RD) = 45.8, 95% CI 2-sided [22.0 to 69.6] — Statistics for the difference were calculated using unadjusted risk differences (BI dose group - Placebo)
Statistical Analysis 6: Comparison: Part II - Placebo (Fed) vs Part II - BI 200 mg Twice Daily, 400 mg Total (Fed); [analysis description as in outcome 1, analysis 5]; Test type: Other; Risk Difference (RD) = 35.2, 95% CI 2-sided [11.3 to 59.2] — Statistics for the difference were calculated using unadjusted risk differences (BI dose group - Placebo)

4. Secondary Outcome: Number of Patients Who Achieved Psoriasis Area Severity Index Score (PASI) 90 at Week 12
Description: Number of patients who achieved Psoriasis Area Severity Index score (PASI) 90 at week 12. The PASI is a tool which provides a numeric scoring for patients overall psoriasis disease state, ranging from 0 to 72. It is a linear combination of percent of surface area of skin that is affected and the severity of erythema, infiltration, and desquamation over four body regions. Higher scores indicating higher severity, while a score of 0 indicates no disease.
  PASI 90 is based on the percent reduction from baseline, generally summarized as a dichotomous outcome based on achieving over an 90% reduction.
  No statistical comparisons were planned or carried out for Part 2 of the trial. Statistical analysis could not be performed for arms with 0 participants reaching PASI 90.
Time Frame: Assesment at week 12 of treatment
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part I - Placebo (Fasted) | Part I - BI 25 mg (Fasted) | Part I - BI 50 mg (Fasted) | Part I - BI 100 mg (Fasted) | Part I - BI 200 mg (Fasted) | Part II - Placebo (Fed) | Part II - BI 400 mg Once Daily (Fed) | Part II - BI 200 mg Twice Daily, 400 mg Total (Fed)
Number analyzed (Participants) | 20 | 40 | 39 | 39 | 40 | 10 | 43 | 42
Participants | 0 | 0 | 2 | 1 | 7 | 0 | 4 | 2
Statistical Analysis 1: Comparison: Part I - Placebo (Fasted) vs Part I - BI 50 mg (Fasted); Test type: Other; p = 0.3028, Chi-squared; Risk Difference (RD) = 5.1, 95% CI 2-sided [-1.8 to 12.1] — Statistics for the difference were calculated using unadjusted risk differences (BI dose group - Placebo)
Statistical Analysis 2: Comparison: Part I - Placebo (Fasted) vs Part I - BI 100 mg (Fasted); Test type: Other; p = 0.4701, Chi-squared; Risk Difference (RD) = 2.6, 95% CI 2-sided [-2.4 to 7.5] — Statistics for the difference were calculated using unadjusted risk differences (BI dose group - Placebo)
Statistical Analysis 3: Comparison: Part I - Placebo (Fasted) vs Part I - BI 200 mg (Fasted); Test type: Other; p = 0.0465, Chi-squared; Risk Difference (RD) = 17.5, 95% CI 2-sided [5.7 to 29.3] — Statistics for the difference were calculated using unadjusted risk differences (BI dose group - Placebo)
Statistical Analysis 4: Comparison: Part II - Placebo (Fed) vs Part II - BI 400 mg Once Daily (Fed); [analysis description as in outcome 1, analysis 5]; Test type: Other; Risk Difference (RD) = 9.3, 95% CI 2-sided [0.6 to 18.0] — Statistics for the difference were calculated using unadjusted risk differences (BI dose group - Placebo)
Statistical Analysis 5: Comparison: Part II - Placebo (Fed) vs Part II - BI 200 mg Twice Daily, 400 mg Total (Fed); [analysis description as in outcome 1, analysis 5]; Test type: Other; Risk Difference (RD) = 4.8, 95% CI 2-sided [-1.7 to 11.2] — Statistics for the difference were calculated using unadjusted risk differences (BI dose group - Placebo)

5. Secondary Outcome: Number of Patients Who Achieved Psoriasis Area Severity Index Score (PASI) 100 at Week 12
Description: Number of patients who achieved Psoriasis Area Severity Index score (PASI) 100 at week 12. The PASI is a tool which provides a numeric scoring for patients overall psoriasis disease state, ranging from 0 to 72. It is a linear combination of percent of surface area of skin that is affected and the severity of erythema, infiltration, and desquamation over four body regions. Higher scores indicating higher severity, while a score of 0 indicates no disease.
  PASI 100 is based on the percent reduction from baseline, generally summarized as a dichotomous outcome based on achieving over an 100% reduction.
  No statistical comparisons were planned or carried out for Part 2 of the trial. Statistical analysis could not be performed for arms with 0 participants reaching PASI 100.
Time Frame: Assesment at week 12 of treatment
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part I - Placebo (Fasted) | Part I - BI 25 mg (Fasted) | Part I - BI 50 mg (Fasted) | Part I - BI 100 mg (Fasted) | Part I - BI 200 mg (Fasted) | Part II - Placebo (Fed) | Part II - BI 400 mg Once Daily (Fed) | Part II - BI 200 mg Twice Daily, 400 mg Total (Fed)
Number analyzed (Participants) | 20 | 40 | 39 | 39 | 40 | 10 | 43 | 42
Participants | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 2
Statistical Analysis 1: Comparison: Part I - Placebo (Fasted) vs Part I - BI 100 mg (Fasted); Test type: Other; p = 0.4701, Chi-squared; Risk Difference (RD) = 2.6, 95% CI 2-sided [-2.4 to 7.5] — Statistics for the difference were calculated using unadjusted risk differences (BI dose group - Placebo)
Statistical Analysis 2: Comparison: Part I - Placebo (Fasted) vs Part I - BI 200 mg (Fasted); Test type: Other; p = 0.3091, Chi-squared; Risk Difference (RD) = 5.0, 95% CI 2-sided [-1.8 to 11.8] — Statistics for the difference were calculated using unadjusted risk differences (BI dose group - Placebo)
Statistical Analysis 3: Comparison: Part II - Placebo (Fed) vs Part II - BI 400 mg Once Daily (Fed); [analysis description as in outcome 1, analysis 5]; Test type: Other; Risk Difference (RD) = 2.3, 95% CI 2-sided [-2.2 to 6.8] — Statistics for the difference were calculated using unadjusted risk differences (BI dose group - Placebo)
Statistical Analysis 4: Comparison: Part II - Placebo (Fed) vs Part II - BI 200 mg Twice Daily, 400 mg Total (Fed); [analysis description as in outcome 1, analysis 5]; Test type: Other; Risk Difference (RD) = 2.4, 95% CI 2-sided [-2.2 to 7.0] — Statistics for the difference were calculated using unadjusted risk differences (BI dose group - Placebo)

6. Secondary Outcome: Number of Patients Who Achieved Psoriasis Area Severity Index Score (PASI) 75 at Weeks 16, 20, and 24
Description: Number of patients who achieved Psoriasis Area Severity Index score (PASI) 75 at weeks 16, 20 and 24. The PASI is a tool which provides a numeric scoring for patients overall psoriasis disease state, ranging from 0 to 72. It is a linear combination of percent of surface area of skin that is affected and the severity of erythema, infiltration, and desquamation over four body regions. Higher scores indicating higher severity, while a score of 0 indicates no disease.
  PASI 75 is based on the percent reduction from baseline, generally summarized as a dichotomous outcome based on achieving over an 75% reduction.
Time Frame: Assesment at week 16, 20 and 24 of treatment
Population: Full Analysis Set (FAS): The FAS includes all patients who received at least 1 dose of trial medication and provided baseline and at least 1 post-randomisation measurement of Psoriasis Area Severity Index (PASI). Subjects with missing data for subsequent visits were included but those entries were imputed as failures. Subjects with missing data for subsequent visits were included but those entries were imputed as failures.
Measure: Count of Participants; unit: Participants
Arm/Group | Part I - Placebo (Fasted) | Part I - BI 25 mg (Fasted) | Part I - BI 50 mg (Fasted) | Part I - BI 100 mg (Fasted) | Part I - BI 200 mg (Fasted)
Number analyzed (Participants) | 20 | 40 | 39 | 39 | 40
Participants
  Week 16 | 0 | 1 | 1 | 5 | 11
  Week 20 | 0 | 2 | 3 | 4 | 13
  Week 24 | 0 | 2 | 4 | 4 | 14
Statistical Analysis 1: Comparison: Part I - Placebo (Fasted) vs Part I - BI 25 mg (Fasted); Test type: Other; p = 0.4758, Chi-squared; Risk Difference (RD) = 2.5, 95% CI 2-sided [-2.3 to 7.3] — Statistics for the difference were calculated using unadjusted risk differences (BI dose group - Placebo)
Statistical Analysis 2: Comparison: Part I - Placebo (Fasted) vs Part I - BI 50 mg (Fasted); Test type: Other; p = 0.4701, Chi-squared; Risk Difference (RD) = 2.6, 95% CI 2-sided [-2.4 to 7.5] — Statistics for the difference were calculated using unadjusted risk differences (BI dose group - Placebo)
Statistical Analysis 3: Comparison: Part I - Placebo (Fasted) vs Part I - BI 100 mg (Fasted); Test type: Other; p = 0.0942, Chi-squared; Risk Difference (RD) = 12.8, 95% CI 2-sided [2.3 to 23.3] — Statistics for the difference were calculated using unadjusted risk differences (BI dose group - Placebo)
Statistical Analysis 4: Comparison: Part I - Placebo (Fasted) vs Part I - BI 200 mg (Fasted); Test type: Other; p = 0.0095, Chi-squared; Risk Difference (RD) = 27.5, 95% CI 2-sided [13.7 to 41.3] — Statistics for the difference were calculated using unadjusted risk differences (BI dose group - Placebo)
Statistical Analysis 5: Comparison: Part I - Placebo (Fasted) vs Part I - BI 25 mg (Fasted); Test type: Other; p = 0.3091, Chi-squared; Risk Difference (RD) = 5.0, 95% CI 2-sided [-1.8 to 11.8] — Statistics for the difference were calculated using unadjusted risk differences (BI dose group - Placebo)
Statistical Analysis 6: Comparison: Part I - Placebo (Fasted) vs Part I - BI 50 mg (Fasted); Test type: Other; p = 0.2030, Chi-squared; Risk Difference (RD) = 7.7, 95% CI 2-sided [-0.7 to 16.1] — Statistics for the difference were calculated using unadjusted risk differences (BI dose group - Placebo)
Statistical Analysis 7: Comparison: Part I - Placebo (Fasted) vs Part I - BI 100 mg (Fasted); Test type: Other; p = 0.1380, Chi-squared; Risk Difference (RD) = 10.3, 95% CI 2-sided [0.7 to 19.8] — Statistics for the difference were calculated using unadjusted risk differences (BI dose group - Placebo)
Statistical Analysis 8: Comparison: Part I - Placebo (Fasted) vs Part I - BI 200 mg (Fasted); Test type: Other; p = 0.0040, Chi-squared; Risk Difference (RD) = 32.5, 95% CI 2-sided [18.0 to 47.0] — Statistics for the difference were calculated using unadjusted risk differences (BI dose group - Placebo)
Statistical Analysis 9: Comparison: Part I - Placebo (Fasted) vs Part I - BI 50 mg (Fasted); Test type: Other; p = 0.1380, Chi-squared; Risk Difference (RD) = 10.3, 95% CI 2-sided [0.7 to 19.8] — Statistics for the difference were calculated using unadjusted risk differences (BI dose group - Placebo)
Statistical Analysis 10: Comparison: Part I - Placebo (Fasted) vs Part I - BI 200 mg (Fasted); Test type: Other; p = 0.0025, Chi-squared; Risk Difference (RD) = 35.0, 95% CI 2-sided [20.2 to 49.8] — Statistics for the difference were calculated using unadjusted risk differences (BI dose group - Placebo)

7. Secondary Outcome: Number of Patients Who Achieved a Static Physician's Global Assessment Score of 'Clear' (sPGA 0) at Week 12
Description: Number of patients who achieved a static Physician's Global Assessment score of 'clear' (sPGA 0) at Week 12. The sPGA used in this trial is a 5 point score ranging from 0 to 4, based on the physician's assessment of the average thickness, erythema, and scaling of all psoriatic lesions. The assessment is considered "static" which refers to the patients disease state at the time of the assessments, without comparison to any of the subject's previous disease states, whether at Baseline or at a previous visit. A lower score indicates less body coverage, with 0 being clear and 1 being almost clear.
  No statistical comparisons were planned or carried out for Part 2 of the trial.
Time Frame: Assesment at week 12 of treatment
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part I - Placebo (Fasted) | Part I - BI 25 mg (Fasted) | Part I - BI 50 mg (Fasted) | Part I - BI 100 mg (Fasted) | Part I - BI 200 mg (Fasted) | Part II - Placebo (Fed) | Part II - BI 400 mg Once Daily (Fed) | Part II - BI 200 mg Twice Daily, 400 mg Total (Fed)
Number analyzed (Participants) | 20 | 40 | 39 | 39 | 40 | 10 | 43 | 42
Participants | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 1
Statistical Analysis 1: Comparison: Part I - Placebo (Fasted) vs Part I - BI 100 mg (Fasted); Test type: Other; p = 0.4701, Chi-squared; Risk Difference (RD) = 2.6, 95% CI 2-sided [-2.4 to 7.5] — Statistics for the difference were calculated using unadjusted risk differences (BI dose group - Placebo)
Statistical Analysis 2: Comparison: Part I - Placebo (Fasted) vs Part I - BI 200 mg (Fasted); Test type: Other; p = 0.3091, Chi-squared; Risk Difference (RD) = 5.0, 95% CI 2-sided [-1.8 to 11.8] — Statistics for the difference were calculated using unadjusted risk differences (BI dose group - Placebo)

8. Secondary Outcome: Number of Patients Who Achieved a Static Physician's Global Assessment Score of 'Clear' or 'Almost Clear' (sPGA 0/1) at Weeks 16, 20, and 24
Description: Number of patients who achieved a static Physician's Global Assessment score of 'clear' or 'almost clear' (sPGA 0/1) at Week 16, 20 and 24. The sPGA used in this trial is a 5 point score ranging from 0 to 4, based on the physician's assessment of the average thickness, erythema, and scaling of all psoriatic lesions. The assessment is considered "static" which refers to the patients disease state at the time of the assessments, without comparison to any of the subject's previous disease states, whether at Baseline or at a previous visit. A lower score indicates less body coverage, with 0 being clear and 1 being almost clear.
Time Frame: Assesment at week 16, 20 and 24 of treatment
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part I - Placebo (Fasted) | Part I - BI 25 mg (Fasted) | Part I - BI 50 mg (Fasted) | Part I - BI 100 mg (Fasted) | Part I - BI 200 mg (Fasted)
Number analyzed (Participants) | 20 | 40 | 39 | 39 | 40
Participants
  Week 16 | 0 | 1 | 2 | 3 | 12
  Week 20 | 0 | 1 | 4 | 2 | 10
  Week 24 | 0 | 1 | 3 | 4 | 13
Statistical Analysis 1: Comparison: Part I - Placebo (Fasted) vs Part I - BI 25 mg (Fasted); Test type: Other; p = 0.4758, Chi-squared; Risk Difference (RD) = 2.5, 95% CI 2-sided [-2.3 to 7.3] — Statistics for the difference were calculated using unadjusted risk differences (BI dose group - Placebo)
Statistical Analysis 2: Comparison: Part I - Placebo (Fasted) vs Part I - BI 50 mg (Fasted); Test type: Other; p = 0.3028, Chi-squared; Risk Difference (RD) = 5.1, 95% CI 2-sided [-1.8 to 12.1] — Statistics for the difference were calculated using unadjusted risk differences (BI dose group - Placebo)
Statistical Analysis 3: Comparison: Part I - Placebo (Fasted) vs Part I - BI 100 mg (Fasted); Test type: Other; p = 0.2030, Chi-squared; Risk Difference (RD) = 7.7, 95% CI 2-sided [-0.7 to 16.1] — Statistics for the difference were calculated using unadjusted risk differences (BI dose group - Placebo)
Statistical Analysis 4: Comparison: Part I - Placebo (Fasted) vs Part I - BI 200 mg (Fasted); Test type: Other; p = 0.0062, Chi-squared; Risk Difference (RD) = 30.0, 95% CI 2-sided [15.8 to 44.2] — Statistics for the difference were calculated using unadjusted risk differences (BI dose group - Placebo)
Statistical Analysis 5: Comparison: Part I - Placebo (Fasted) vs Part I - BI 50 mg (Fasted); Test type: Other; p = 0.1380, Chi-squared; Risk Difference (RD) = 10.3, 95% CI 2-sided [0.7 to 19.8] — Statistics for the difference were calculated using unadjusted risk differences (BI dose group - Placebo)
Statistical Analysis 6: Comparison: Part I - Placebo (Fasted) vs Part I - BI 100 mg (Fasted); Test type: Other; p = 0.3028, Chi-squared; Risk Difference (RD) = 5.1, 95% CI 2-sided [-1.8 to 12.1] — Statistics for the difference were calculated using unadjusted risk differences (BI dose group - Placebo)
Statistical Analysis 7: Comparison: Part I - Placebo (Fasted) vs Part I - BI 200 mg (Fasted); Test type: Other; p = 0.0143, Chi-squared; Risk Difference (RD) = 25.0, 95% CI 2-sided [11.6 to 38.4] — Statistics for the difference were calculated using unadjusted risk differences (BI dose group - Placebo)
Statistical Analysis 8: Comparison: Part I - Placebo (Fasted) vs Part I - BI 50 mg (Fasted); Test type: Other; p = 0.2030, Chi-squared; Risk Difference (RD) = 7.7, 95% CI 2-sided [-0.7 to 16.1] — Statistics for the difference were calculated using unadjusted risk differences (BI dose group - Placebo)
Statistical Analysis 9: Comparison: Part I - Placebo (Fasted) vs Part I - BI 100 mg (Fasted); Test type: Other; p = 0.1380, Chi-squared; Risk Difference (RD) = 10.3, 95% CI 2-sided [0.7 to 19.8] — Statistics for the difference were calculated using unadjusted risk differences (BI dose group - Placebo)
Statistical Analysis 10: Comparison: Part I - Placebo (Fasted) vs Part I - BI 200 mg (Fasted); Test type: Other; p = 0.0040, Chi-squared; Risk Difference (RD) = 32.5, 95% CI 2-sided [18.0 to 47.0] — Statistics for the difference were calculated using unadjusted risk differences (BI dose group - Placebo)

9. Secondary Outcome: Overall Change From Baseline in Psoriasis Symptoms Evaluated Using the Total Score of the Psoriasis Symptoms Scale (PSS) at Week 12
Description: Overall change from baseline in psoriasis symptoms evaluated using the total score of the Psoriasis Symptoms Scale (PSS) at Week 12. The PSS is a four-item patient-reported outcome (PRO) instrument that assesses the severity of psoriasis symptoms in patients with moderate to severe psoriasis. The symptoms included are: pain, redness, itching and burning from psoriasis.
  Current symptom severity is assessed for a 24 hour recall period using a 5-point verbal rating scale, the PSS score ranges from 0 (none) to 4 (very severe). The symptom scores are added to an unweighted total score (range: 0 to 16).
  Presented 'Mean' values are actually 'Adjusted Mean'. No hypothesis testing was planned or carried out for Part II.
Time Frame: Assesment at week 12 of treatment
Population: Full Analysis Set (FAS): All patients who received at least 1 dose of trial medication and provided a baseline and at least 1 postrandomisation measurement of PASI. Only participants with non-missing values are reported.
Measure: Mean (Standard Error); unit: Total score
Arm/Group | Part I - Placebo (Fasted) | Part I - BI 25 mg (Fasted) | Part I - BI 50 mg (Fasted) | Part I - BI 100 mg (Fasted) | Part I - BI 200 mg (Fasted) | Part II - Placebo (Fed) | Part II - BI 400 mg Once Daily (Fed) | Part II - BI 200 mg Twice Daily, 400 mg Total (Fed)
Number analyzed (Participants) | 20 | 40 | 38 | 38 | 40 | 10 | 43 | 42
Total score | -0.4 (1.0) | 0.1 (0.7) | 0.2 (0.7) | 2.3 (0.7) | 3.6 (0.7) | 0.3 (1.2) | 3.4 (0.6) | 3.3 (0.6)
Statistical Analysis 1: Comparison: Part I - Placebo (Fasted) vs Part I - BI 25 mg (Fasted); Test type: Other; p = 0.7008, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Adjusted mean = 0.5, 95% CI 2-sided [-1.9 to 2.8], Standard Error of Mean 1.2 — MMRM model included treatment, visit and treatment by visit as fixed effects, baseline PSS score and baseline PSS by visit as covariates, patient as a random effect, and an unstructured covariance structure for within patient variation
Statistical Analysis 2: Comparison: Part I - Placebo (Fasted) vs Part I - BI 50 mg (Fasted); Test type: Other; p = 0.6268, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Adjusted mean = 0.6, 95% CI 2-sided [-1.8 to 3.0], Standard Error of Mean 1.2 — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 3: Comparison: Part I - Placebo (Fasted) vs Part I - BI 100 mg (Fasted); Test type: Other; p = 0.0266, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Adjusted mean = 2.7, 95% CI 2-sided [0.3 to 5.1], Standard Error of Mean 1.2 — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 4: Comparison: Part I - Placebo (Fasted) vs Part I - BI 200 mg (Fasted); Test type: Other; p = 0.0009, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Adjusted mean = 4.0, 95% CI 2-sided [1.7 to 6.3], Standard Error of Mean 1.2 — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 5: Comparison: Part II - Placebo (Fed) vs Part II - BI 400 mg Once Daily (Fed); Test type: Other; Adjusted mean = 3.1, 95% CI 2-sided [0.4 to 5.8], Standard Error of Mean 1.4 — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 6: Comparison: Part II - Placebo (Fed) vs Part II - BI 200 mg Twice Daily, 400 mg Total (Fed); Test type: Other; Adjusted mean = 3.1, 95% CI 2-sided [0.4 to 5.8], Standard Error of Mean 1.4 — [estimate comment as in outcome 9, analysis 1]

10. Secondary Outcome: Number of Patients Who Achieved a Dermatology Life Quality Index Score of 'no Effect on Patient's Life' (DLQI 0/1) at Week 12
Description: Number of patients who achieved a Dermatology Life Quality Index score of 'no effect on patient's life' (DLQI 0/1) at Week 12. The DLQI is a subject-administered, ten-question, quality of life questionnaire covering 6 domains including symptoms and feelings, daily activities, leisure, work and school, personal relationships and treatment. Item scores range from 0 (not relevant/not at all) to 3 (very much). Question 7 is a "yes"/ "no" question where "yes" is scored as 3. DLQI total score is calculated by summing the scores of each question resulting in a range of 0 to 30 where 0-1 = no effect on subject's life, 2-5 = small effect, 6-10 = moderate effect, 11-20 = very large effect, and 21-30 = extremely large effect on subject's life. The higher the score, the more the quality of life is impaired. A 4-point change from baseline is considered a clinically important difference. No hypothesis testing was planned or carried out for Part II.
Time Frame: Assesment at week 12 of treatment
Population: Full Analysis Set (FAS): All patients who received at least 1 dose of trial medication and provided a baseline and at least 1 postrandomisation measurement of PASI. Subjects with missing data for subsequent visits were included but those entries were imputed as failures.
Measure: Count of Participants; unit: Participants
Arm/Group | Part I - Placebo (Fasted) | Part I - BI 25 mg (Fasted) | Part I - BI 50 mg (Fasted) | Part I - BI 100 mg (Fasted) | Part I - BI 200 mg (Fasted) | Part II - Placebo (Fed) | Part II - BI 400 mg Once Daily (Fed) | Part II - BI 200 mg Twice Daily, 400 mg Total (Fed)
Number analyzed (Participants) | 20 | 40 | 39 | 39 | 40 | 10 | 43 | 42
Participants | 1 | 3 | 3 | 3 | 8 | 2 | 12 | 11
Statistical Analysis 1: Comparison: Part I - Placebo (Fasted) vs Part I - BI 25 mg (Fasted); Test type: Other; p = 0.7144, Chi-squared; Risk Difference (RD) = 2.5, 95% CI 2-sided [-10.1 to 15.1] — Statistics for the difference were calculated using unadjusted risk differences (BI dose group - Placebo)
Statistical Analysis 2: Comparison: Part I - Placebo (Fasted) vs Part I - BI 50 mg (Fasted); Test type: Other; p = 0.6970, Chi-squared; Risk Difference (RD) = 2.7, 95% CI 2-sided [-10.0 to 15.4] — Statistics for the difference were calculated using unadjusted risk differences (BI dose group - Placebo)
Statistical Analysis 3: Comparison: Part I - Placebo (Fasted) vs Part I - BI 100 mg (Fasted); Test type: Other; p = 0.6970, Chi-squared; Risk Difference (RD) = 2.7, 95% CI 2-sided [-10.0 to 15.4] — Statistics for the difference were calculated using unadjusted risk differences (BI dose group - Placebo)
Statistical Analysis 4: Comparison: Part I - Placebo (Fasted) vs Part I - BI 200 mg (Fasted); Test type: Other; p = 0.1250, Chi-squared; Risk Difference (RD) = 15.0, 95% CI 2-sided [-0.6 to 30.6] — Statistics for the difference were calculated using unadjusted risk differences (BI dose group - Placebo)
Statistical Analysis 5: Comparison: Part II - Placebo (Fed) vs Part II - BI 400 mg Once Daily (Fed); [analysis description as in outcome 1, analysis 5]; Test type: Other; Risk Difference (RD) = 7.9, 95% CI 2-sided [-20.3 to 36.1] — Statistics for the difference were calculated using unadjusted risk differences (BI dose group - Placebo)
Statistical Analysis 6: Comparison: Part II - Placebo (Fed) vs Part II - BI 200 mg Twice Daily, 400 mg Total (Fed); [analysis description as in outcome 1, analysis 5]; Test type: Other; Risk Difference (RD) = 6.2, 95% CI 2-sided [-21.9 to 34.3] — Statistics for the difference were calculated using unadjusted risk differences (BI dose group - Placebo)

ADVERSE EVENTS:
Time Frame: Part I - Period 1: start till the end of treatment in period 1 (week 12) + 7 days residual effect period, up to 13 weeks. Part I - Period 1 and 2 only: start till the end of treatment (week 24) + 7 days residual effect period, up to 25 weeks. Part II: start till the end of treatment (week 12) + 7 days residual effect period, up to 13 weeks. All-cause mortality: start of treatment till the end of treatment + 4 weeks of follow up, up to 28 weeks for Part I and up to 16 weeks for part II.
Description: Treated Set (TS): The TS includes all randomized patients who received at least 1 dose of trial medication and is based on the actual treatment received at randomization visit and week 12 visit, if applicable.
Groups:
- Part I - Period 1 - Fasted: Placebo: Part I - Period 1 - fasted: Placebo matching BI 730357 taken orally daily as a film-coated tablet in the morning while fasted. Participants in this arm only participated in period 1 and did not enter period 2.
- Part I - Period 1 - Fasted: BI 25 mg: Part I - Period 1 - fasted: 25 milligram (mg) BI 730357 taken orally daily as a film-coated tablet in the morning while fasted. Participants in this arm only participated in period 1 and did not enter period 2.
- Part I - Period 1 - Fasted: BI 50 mg: Part I - Period 1 - fasted: 50 milligram (mg) BI 730357 taken orally daily as a film-coated tablet in the morning while fasted. Participants in this arm only participated in period 1 and did not enter period 2.
- Part I - Period 1 - Fasted: BI 100 mg: Part I - Period 1 - fasted: 100 milligram (mg) BI 730357 taken orally daily as a film-coated tablet in the morning while fasted. Participants in this arm only participated in period 1 and did not enter period 2.
- Part I - Period 1 - Fasted: BI 200 mg: Part I - Period 1 - fasted: 200 milligram (mg) BI 730357 taken orally daily as a film-coated tablet in the morning while fasted. Participants in this arm only participated in period 1 and did not enter period 2.
- Part I - Period 1 and 2 - Fasted: Placebo - BI 200 mg: Part I - Period 1 and 2 - fasted: Placebo participants in period who failed to achieve a PASI 75 response at Week 12 and were switched to a 200 mg dose in period 2.
- Part I - Period 1 and 2 - Fasted: BI 25 mg - BI 25 mg: Part I - Period 1 and 2 - fasted: 25 milligram (mg) BI 730357 taken orally daily as a film-coated tablet in the morning while fasted in period 1. Participants who achieved a PASI 50 response at Week 12 and stayed on a 25 mg dose in period 2.
- Part I - Period 1 and 2 - Fasted: BI 25 mg - BI 50 mg: Part I - Period 1 and 2 - fasted: Participants assigned 25 milligram (mg) BI 730357 in period 1 (taken orally daily as a film-coated tablet in the morning while fasted) who failed to achieve a PASI 50 response at Week 12 and were switched to a 50 mg dose in period 2.
- Part I - Period 1 and 2 - Fasted: BI 50 mg - BI 50 mg: Part I - Period 1 and 2 - fasted: 50 milligram (mg) BI 730357 taken orally daily as a film-coated tablet in the morning while fasted in period 1. Participants who achieved a PASI 50 response at Week 12 and stayed on a 50 mg dose in period 2.
- Part I - Period 1 and 2 - Fasted: BI 50 mg - BI 100 mg: Part I - Period 1 and 2 - fasted: Participants assigned 50 milligram (mg) BI 730357 in period 1 (taken orally daily as a film-coated tablet in the morning while fasted) who failed to achieve a PASI 50 response at Week 12 and were switched to a 100 mg dose in period 2.
- Part I - Period 1 and 2 - Fasted: BI 100 mg - BI 100 mg: Part I - Period 1 and 2 - fasted: 100 milligram (mg) BI 730357 taken orally daily as a film-coated tablet in the morning while fasted in period 1. Participants who achieved a PASI 50 response at Week 12 and stayed on a 100 mg dose in period 2.
- Part I - Period 1 and 2 - Fasted: BI 100 mg - BI 200 mg: Part I - Period 1 and 2 - fasted: Participants assigned 100 milligram (mg) BI 730357 in period 1 (taken orally daily as a film-coated tablet in the morning while fasted) who failed to achieve a PASI 50 response at Week 12 and were switched to a 200 mg dose in period 2.
- Part I - Period 1 and 2 - Fasted: BI 200 mg - BI 200 mg: Part I - Period 1 and 2 - fasted: Participants assigned 200 milligram (mg) BI 730357 in period 1 (taken orally daily as a film-coated tablet in the morning while fasted) who remained on the 200 mg throughout period 1 and 2.
Arm/Group | Part I - Period 1 - Fasted: Placebo | Part I - Period 1 - Fasted: BI 25 mg | Part I - Period 1 - Fasted: BI 50 mg | Part I - Period 1 - Fasted: BI 100 mg | Part I - Period 1 - Fasted: BI 200 mg | Part I - Period 1 and 2 - Fasted: Placebo - BI 200 mg | Part I - Period 1 and 2 - Fasted: BI 25 mg - BI 25 mg | Part I - Period 1 and 2 - Fasted: BI 25 mg - BI 50 mg | Part I - Period 1 and 2 - Fasted: BI 50 mg - BI 50 mg | Part I - Period 1 and 2 - Fasted: BI 50 mg - BI 100 mg | Part I - Period 1 and 2 - Fasted: BI 100 mg - BI 100 mg | Part I - Period 1 and 2 - Fasted: BI 100 mg - BI 200 mg | Part I - Period 1 and 2 - Fasted: BI 200 mg - BI 200 mg | Part II - Placebo (Fed) | Part II - BI 400 mg Once Daily (Fed) | Part II - BI 200 mg Twice Daily, 400 mg Total (Fed)
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/3 | 0/8 | 0/6 | 0/3 | 0/15 | 0/2 | 0/35 | 0/10 | 0/21 | 0/8 | 0/25 | 0/37 | 0/10 | 0/44 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/3 | 0/8 | 0/6 | 0/3 | 0/15 | 0/2 | 2/35 | 0/10 | 1/21 | 0/8 | 0/25 | 0/37 | 0/10 | 0/44 | 0/42
Other Adverse Events (participants affected / at risk) | 4/5 | 2/3 | 2/8 | 2/6 | 3/3 | 9/15 | 1/2 | 15/35 | 7/10 | 13/21 | 7/8 | 12/25 | 18/37 | 5/10 | 9/44 | 8/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part I - Period 1 - Fasted: Placebo (N=5) | Part I - Period 1 - Fasted: BI 25 mg (N=3) | Part I - Period 1 - Fasted: BI 50 mg (N=8) | Part I - Period 1 - Fasted: BI 100 mg (N=6) | Part I - Period 1 - Fasted: BI 200 mg (N=3) | Part I - Period 1 and 2 - Fasted: Placebo - BI 200 mg (N=15) | Part I - Period 1 and 2 - Fasted: BI 25 mg - BI 25 mg (N=2) | Part I - Period 1 and 2 - Fasted: BI 25 mg - BI 50 mg (N=35) | Part I - Period 1 and 2 - Fasted: BI 50 mg - BI 50 mg (N=10) | Part I - Period 1 and 2 - Fasted: BI 50 mg - BI 100 mg (N=21) | Part I - Period 1 and 2 - Fasted: BI 100 mg - BI 100 mg (N=8) | Part I - Period 1 and 2 - Fasted: BI 100 mg - BI 200 mg (N=25) | Part I - Period 1 and 2 - Fasted: BI 200 mg - BI 200 mg (N=37) | Part II - Placebo (Fed) (N=10) | Part II - BI 400 mg Once Daily (Fed) (N=44) | Part II - BI 200 mg Twice Daily, 400 mg Total (Fed) (N=42)
Comminuted fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part I - Period 1 - Fasted: Placebo (N=5) | Part I - Period 1 - Fasted: BI 25 mg (N=3) | Part I - Period 1 - Fasted: BI 50 mg (N=8) | Part I - Period 1 - Fasted: BI 100 mg (N=6) | Part I - Period 1 - Fasted: BI 200 mg (N=3) | Part I - Period 1 and 2 - Fasted: Placebo - BI 200 mg (N=15) | Part I - Period 1 and 2 - Fasted: BI 25 mg - BI 25 mg (N=2) | Part I - Period 1 and 2 - Fasted: BI 25 mg - BI 50 mg (N=35) | Part I - Period 1 and 2 - Fasted: BI 50 mg - BI 50 mg (N=10) | Part I - Period 1 and 2 - Fasted: BI 50 mg - BI 100 mg (N=21) | Part I - Period 1 and 2 - Fasted: BI 100 mg - BI 100 mg (N=8) | Part I - Period 1 and 2 - Fasted: BI 100 mg - BI 200 mg (N=25) | Part I - Period 1 and 2 - Fasted: BI 200 mg - BI 200 mg (N=37) | Part II - Placebo (Fed) (N=10) | Part II - BI 400 mg Once Daily (Fed) (N=44) | Part II - BI 200 mg Twice Daily, 400 mg Total (Fed) (N=42)
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Photophobia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 1
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 3
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bacteriuria (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Chlamydial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hand-foot-and-mouth disease (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lyme disease (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 3 | 1 | 2 | 3 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 3 | 1 | 1 | 2 | 4 | 1 | 2 | 7 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 2 | 0 | 2 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nail avulsion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Electrocardiogram ST segment depression (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0
Liver function test increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0
Occult blood positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pancreatic enzymes increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Prothrombin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 1
Migraine (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Uterine spasm (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intertrigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0 | 0 | 2 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0
Defect conduction intraventricular (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2020-08-24): https://cdn.clinicaltrials.gov/large-docs/99/NCT03635099/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-12): https://cdn.clinicaltrials.gov/large-docs/99/NCT03635099/SAP_001.pdf